CLINICAL TRIAL: NCT00794742
Title: Analyzing the Antimicrobial Resistance Profile of Bacterial Isolates Obtained From Severely Burned Patients
Brief Title: Antimicrobial Resistance of Bacteria in Burn Patients
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: TTUHSC-L09-014
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Burns
Keywords: Burn; Antimicrobial; Bacteria; Resistance; Biofilm; Pathogen
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacterial isolates of infected burn wounds
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Burn Wounds: Patients with burn wounds

SUMMARY:
The purpose of this study is to test the resistance of pathogenic bacteria in infected tissues of burn patients to various antimicrobials and enzyme debriders.

DETAILED DESCRIPTION:
Bacteria that is present in infected burn wounds will be isolated and identified. The isolates will be tested for resistance to commercially available antimicrobials.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any age
* Have open, unhealed wounds(s) that will be cultured per standard of care
* Subject or authorized representative provide informed consent

Exclusion Criteria:

* Informed consent not provided or able to be obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with open,unhealed,burn wounds
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Types of bacteria | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: John Griswold, M.D., Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- University Medical Center, Lubbock, Texas, United States